CLINICAL TRIAL: NCT00802516
Title: Effects of Long-term Daily Consumption of Plant Sterol or Stanol Esters in Statin-treated Patients
Brief Title: Long Term Effects of Plant Sterol and Stanol Esters
Acronym: LTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Jogchem Plat PhD, Maastricht UMC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MEC03-046.3
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2008-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. placebo (Placebo Comparator): placebo margarine
  Interventions: Dietary Supplement: No intervention
- 2. stanol ester (Experimental): margarine with plant stanol ester
  Interventions: Dietary Supplement: stanol ester
- 3. sterol ester (Experimental): margarine with plant sterol ester
  Interventions: Dietary Supplement: sterol ester

INTERVENTIONS:
Dietary Supplement: stanol ester — enriched margarine
  Arms: 2. stanol ester
Dietary Supplement: sterol ester — enriched margarine
  Arms: 3. sterol ester
Dietary Supplement: No intervention — placebo margarine
  Arms: 1. placebo

SUMMARY:
BACKGROUND Plant sterols and stanols are compounds that are structurally related to cholesterol, which decrease intestinal cholesterol absorption and consequently serum LDL cholesterol concentrations by 10-14%. Nowadays plant sterols and stanols are widely available incorporated in food products like margarines and yogurts and are presented as functional foods.

Whether the cholesterol lowering effects of plant sterols and stanols also favorably affect endothelial function in humans is currently unknown. Apart from their cholesterol lowering effects, plant sterols and stanols might have other effects like effects on red blood cell properties, cognitive performance and antioxidant status. Especially to evaluate effects on this type of parameters long-term daily consumption of plant sterols and stanols is necessary. These questions will be answered in statin treated patients since functional foods enriched with plant sterol and stanol esters have been recommended for statin-users as an "add on" therapy. This may ultimately lead to a lower dose of statins or an increased number of patients that reach the target for LDL-cholesterol reduction.

AIM The major objective of the present proposal is to examine the effects of a long-term consumption of plant sterols and stanols on the endothelial function of the vessel wall in statin-treated patients.

STUDY DESIGN Subjects: The subjects will be recruited among men and women in Maastricht and surroundings, aged between 18 and 70 years. Participation will be on voluntary basis. People who are willing to participate will be invited for two screening visits.

Experimental design: The present study is a double-blind, randomized parallel intervention trial with 60 statin-treated subjects, in which the metabolic effects of a long term (90 weeks) consumption of plant sterols and stanols (2.5 g/day) will be studied. After a run-in period of 5 weeks the subjects will be randomly divided into three groups of 20 subjects each. One group will continue with the control margarine without added plant sterols and stanols, one group will use a plant sterol margarine and the last group will use a plant stanol margarine for 85 weeks. The major endpoint will be endothelial function of the vessel wall, and in addition various parameters related to lipids and lipoprotein metabolism, erythrocyte characteristics and cognitive performance will be measured.

Risk for subjects The margarines containing the plant sterols and stanols are safe and palatable. Venipunctures and other (non-invasive) measurements are carried out by skilled persons and not of any risk. A subject will spend approximately 1 hour a month in participating in the studies.

ELIGIBILITY:
Inclusion Criteria:

* Statin-treatment
* Stable dietary habits

Exclusion Criteria:

* Active cardiovascular disease like congestive heart failure or recent (< 6 months) event (acute myocardial infarction, CVA)
* Impairment of renal function, as evidenced by increased serum creatinine > 150 mcmol/L
* Hepatic diseases as manifested by ALT, AST, GGT, total bilirubin or ALP > 2 times the upper limit of normal
* Severe medical conditions that might interfere with the study such as epilepsy, asthma, and rheumatoid arthritis.
* Use of medication such as corticosteroids, diuretics or lipid lowering medication other than statins
* Unstable body weight (weight gain or loss >3 kg in the past three months)
* Abnormal hematological profile
* Quetelet-index > 32 kg/m2
* Diastolic blood pressure > 100 mm Hg or systolic > 160 mm Hg
* Abuse of drugs and/or alcohol
* Use of sterol or stanol ester products within the previous 30 days
* Participation in another study within 1 months prior to the screening visit
* Pregnant women or women with child-wish within the duration of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-06; Primary Completion 2005-01 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
the endothelial function of the vessel wall in statin-treated patients. | 85 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jogchem Plat, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University, Maastricht, Netherlands